CLINICAL TRIAL: NCT03560180
Title: Early Diagnosis of Anastomotic Leakage After Colorectal Surgery: a Prospective Observational Validation Study of the Dutch Leakage Score, Serum Procalcitonin and Serum CRP: the Italian ColoRectal Anastomotic Leakage (iCRAL) Study Group.
Brief Title: Early Diagnosis of Anastomotic Leakage After Colorectal Surgery: Italian ColoRectal Anastomotic Leakage Study Group.
Acronym: iCral
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale C & G Mazzoni (Other)
Responsible Party: Principal Investigator, Marco Catarci, Director, General Surgery Unit, Ospedale C & G Mazzoni
Other Study IDs: 01/2017
Record Dates: First submitted 2018-06-04; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Anastomotic Leak; Colorectal Surgery
Keywords: Anastomotic Leak; Colorectal Surgery
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dutch score — leakage score (DUtch LeaKage, DULK), that consider several items (fever, heart rate, respiratory rate, urinary production, mental status, clinical conditions, signs of ileus, gastric retention, fascial dehiscence, abdominal pain, wound pain, leukocytosis, CRP, increase of urea or creatinine and nutrition status), to give a score
  Other Names: Dulk score, Anastomotic Leakage Clinical score
Diagnostic Test: Serum C-reactive Protein — see study protocol
Diagnostic Test: serum Procalcitonin — see study protocol

SUMMARY:
Prospective evaluation of early diagnosis of anastomotic leak after colorectal resection through evaluation of Dutch leakage score, serum C-reactive protein and serum Procalcitonin

DETAILED DESCRIPTION:
BACKGROUND

Anastomotic leakage is a dreaded major complication after colorectal surgery. The overall incidence of anastomotic dehiscence and subsequent leaks is 2 to 7 percent when performed by experienced surgeons. The lowest leak rates are found with ileocolic anastomoses (1 to 3 percent) and the highest occur with coloanal anastomosis (10 to 20 percent). Leaks usually become apparent between five and seven days postoperatively. Almost half of all leaks occur after the patient has been discharged, and up to 12 percent occur after postoperative day 30. Late leaks often present insidiously with low-grade fever, prolonged ileus, and nonspecific symptoms attributable to other postoperative infectious complications. Small, contained leaks present later in the clinical course and may be difficult to distinguish from postoperative abscesses by radiologic imaging, making the diagnosis uncertain and underreported.

There is no uniform definition of an anastomotic dehiscence and leak. In a review of 97 studies, as an example, 56 different definitions of an anastomotic leak were used. The majority of reports define an anastomotic leak using clinical signs, radiographic findings, and intraoperative findings. The clinical signs include: Pain, Fever, Tachycardia, Peritonitis, Feculent drainage, Purulent drainage. The radiographic signs include: Fluid collections, Gas containing collections. The intraoperative findings include: Gross enteric spillage, Anastomotic disruption.

Risk factors for a dehiscence and leak are classified according to the site of the anastomosis (extraperitoneal or intraperitoneal). A prospective review of 1598 patients undergoing 1639 anastomotic procedures for benign or malignant colorectal disease found a significantly increased risk of anastomotic leak with extraperitoneal compared with intraperitoneal anastomoses (6.6 versus 1.5 percent; 2.4 percent overall).

Major risk factors for an extraperitoneal anastomotic leak include: The distance of the anastomosis from the anal verge (Patients with a low anterior resection and an anastomosis within 5 cm from the anal verge are the highest risk group for an anastomotic leak), Anastomotic ischemia, Male gender, Obesity.

Major risk factors for an intraperitoneal anastomotic leak include: American Society of Anesthesiologists (ASA) score Grade III to V, Emergent surgery, Prolonged operative time, Hand-sewn ileocolic anastomosis.

Controversial, inconclusive, or pertinent negative associations between the following variables and an anastomotic leak have been reported: Neoadjuvant radiation therapy, Drains, Protective stoma, Hand-sewn colorectal anastomosis, Laparoscopic procedure, Mechanical bowel preparation, Nutritional status, Perioperative corticosteroids.

Early diagnosis is crucial to treat patients limiting the related mortality. For this reason several clinical items were proposed in literature to detect anastomotic leakage as soon as possible: fever, pain, tachycardia, peritoneal, purulent or faecal drain, and dynamic ileus. Moreover, also laboratory markers were proposed, such as leukocytosis, serum procalcitonin (PCT) and C-Reactive Protein (CRP). Finally, in 2009 den Dulk et al. proposed a leakage score (DUtch LeaKage, DULK), that consider several items (fever, heart rate, respiratory rate, urinary production, mental status, clinical conditions, signs of ileus, gastric retention, fascial dehiscence, abdominal pain, wound pain, leukocytosis, CRP, increase of urea or creatinine and nutrition status), to give a score, based on which is chosen a therapeutic strategy.

Therefore, we planned this study to prospectively evaluate anastomotic leakage rate after colorectal resections, trying to give a definite answer to the need for clear risk factors, and testing the diagnostic yeald of DULK score and laboratory markers.

METHODS Prospective enrollment from September 2017 to September 2018 in 19 Italian surgical centers. All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after having provided a written informed consent. A total of 1,131 patients is expected based on a mean of 55 cases/year per center.

Outcome measures

1. Preoperative risk factors of anastomotic leakage (age, gender, obesity, state of nutrition, diabetes, cardiovascular, renal failure, inflammatory bowel disease, ASA class I-II vs III)
2. Operative parameters (approach, procedure, anastomotic technique, time of operation, pTNM stage)
3. Leukocyte count, serum CRP, serum procalcitonin and DULK score assessment in 2nd and 3rd postoperative day. Minor and major complications according to Clavien-Dindo classification
4. Anastomotic leakage rate
5. Morbidity-Mortality rates
6. Length of postoperative hospital stay

Recorded data and follow-up Potential patient-specific and intraoperative risk factors will be recorded: gender, body mass index, nutritional status according to the Mini Nutritional Assessment short-form, surgical indication (cancer, polyps, chronic inflammatory bowel disease, diverticular disease), preoperative albuminemia, use of steroids, renal failure and dialysis, preoperative leukocyte count, CRP, PCT cardiovascular or respiratory disease, American Society of Anesthesia score, bowel preparation (decision made by operating surgeon), laparoscopy or laparotomy, level of anastomosis and technique (mechanical or hand-sewn, intra- or extra-corporeal), operative time, presence of drainage, surgeon and perioperative blood transfusion(s). During the postoperative period, patients will be examined by the attending surgeon daily. Fever (central temperature > 38 °C), pulse, abdominal signs, bowel movements, volume and aspect of drainage (if present) will be recorded daily. Leucocyte count, CRP, PCT and Dulk score will be measured in the evening before the operation (in addition to albuminemia) and on postoperative days 2, 3, and 6 (optional). The attending surgeon will make any decision for complementary exams and imaging according to his own criteria. The rate of any complication will be calculated and graded according to Clavien-Dindo including all leaks (independently of clinical significance), wound infection, pneumonia, central line infection, urinary tract infection. Urinary tract infection will be diagnosed on the basis of positive urine culture with bacterial count. Central line infection will be diagnosed on the basis of positive blood culture. Superficial and deep incisional infections will be diagnosed according to the definitions of the Centers for Disease Control and Prevention and a culture will be performed. Pneumonia will be diagnosed on the basis of clinical symptoms, and physical and radiological examinations. The surgeons will be blinded to the results of the CRP and PCT assays. Patients will be followed-up in the outpatient clinic up to 6 weeks after discharge from the hospital.

Main outcome is anastomotic dehiscence (intended as any deviation from the planned postoperative course related to the anastomosis, or presence of pus or enteric contents within the drains, presence of abdominal or pelvic collection in the area of the anastomosis on postoperative CT scan, performed at the discretion of the attending surgeon, leakage of contrast through the anastomosis during enema or evident anastomotic dehiscence at reoperation for postoperative peritonitis). Thus, all detected leaks will be considered independently of clinical significance. No imaging will be performed routinely in order to search for leakage.

Secondary outcomes are morbidity and mortality rates, and postoperative length of stay. All data will be prospectively recorded into CRF and transmitted to the coordinating center on a monthly basis. Thereafter, all data will be incorporated into a spreadsheet (MS Excel), checking for any discrepancy, that will be addressed and solved through strict cooperation between chief investigator, data manager and participating center.

Statistical Analysis Quantitative values will be expressed as mean ± standard deviation, median and range; categorical data with percentage frequencies. Mean values of duration of stay will be compared according to the presence or absence of fistulas using Student's two-sided t test (allowing for heterogeneity of variances) or with a non-parametric Mann-Whitney test. Mean values of DULK score, CRP and PCT levels will also be compared using Student's two-sided t test (allowing for heterogeneity of variances) or with a non-parametric Mann-Whitney test. Both univariate analysis and multivariate analysis will be performed to assess risk factors for leakage and overall complications. The odds ratio (OR) will be presented followed by its 95% confidence interval (95% CI). Areas under the receiver-operating characteristics (ROC) curve will be calculated. For all statistical tests the significant level is fixed at p < .05. Multivariate analysis will be performed using logistic models. Statistical analyses will be carried out using STATA software (Stata Corp. College Station, Texas, USA).

Sample size Considering that the ASA grade (I and II vs. III) is mostly significant among risk factors for anastomotic dehiscence, an estimation of the OR for anastomotic dehiscence and ASA grade is equal to 5.6; assuming a confidence interval for the estimation of the OR at 95% and a maximum error equal to 0.04, the required sample size is n=1,062 (about 885 and 177 cases expected in ASA I-II and ASA III, respectively).

ELIGIBILITY:
Inclusion Criteria:

1. Patients submitted to laparoscopic/robotic/open/converted ileo-colo-rectal resection with anastomosis (both intra- and/or extra-corporeal), including planned Hartmann's reversals.
2. American Society of Anesthesiologists' (ASA) class I, II or III
3. Elective surgery
4. Patients' written acceptance to be included in the study.

Exclusion Criteria:

1. American Society of Anesthesiologists' (ASA) class IV-V
2. Patients with stoma before or at operation
3. Simple stoma closure
4. Transanal procedure
5. Pregnancy
6. Ongoing infection prior to surgery
7. Hyperthermic intraperitoneal chemotherapy for carcinomatosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective enrollment from September 2017 to September 2018 in 19 Italian surgical centers. All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after having provided a written informed consent.
Sampling Method: Probability Sample
Enrollment: 1131 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leakage | 60 days after operation
  Main outcome is anastomotic dehiscence (intended as any deviation from the planned postoperative course related to the anastomosis, or presence of pus or enteric contents within the drains, presence of abdominal or pelvic collection in the area of the anastomosis on postoperative CT scan, performed at the discretion of the attending surgeon, leakage of contrast through the anastomosis during enema or evident anastomotic dehiscence at reoperation for postoperative peritonitis). Thus, all detected leaks will be considered independently of clinical significance. No imaging will be performed routinely in order to search for leakage.

SECONDARY OUTCOMES:
Operative mortality rates | 60 days after operation
  death due to any cause
Operative morbidity rates | 60 days after operation
  Operative morbidity rates, graded according to Clavien-Dindo classification
Postoperative length of stay | 60 days after operation
  postoperative length of stay expressed in day(s)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Catarci, MD, Study Director — ASUR Marche
Locations (18):
- Italy (18):
  - UOC Chirurgia Generale - Jesi - AV5 - ASUR Marche, Iesi, AN
  - UOC Chirurgia Generale - Ospedale Montichiari (BS) - ASST Spedali Civili di Brescia, Brescia, BS
  - Clinica Chirurgica, Università di Brescia - UOC Chirurgia Generale 3, ASST Spedali Civili di Brescia - Brescia, Brescia, BS
  - S.C. Chirurgia Generale e Oncologica - Azienda Ospedaliera S. Croce e Carle - Cuneo, Italia, Cuneo, CN
  - UOC di Chirurgia Addominale IRCCS Casa Sollievo della Sofferenza - San Giovanni Rotondo - Foggia, San Giovanni Rotondo, FG
  - UOC Chirurgia Generale e Oncologica - Ospedale S. Stefano - Prato (FI) - ASL Toscana Centro, Prato, FI
  - UOC Chirurgia Generale ad Indirizzo Oncologico - IRCCS San Martino IST - Genova, Genova, GE
  - SOC Chirurgia Generale, Oncologica e Vascolare - Azienda Ospedaliera Marche Nord - Pesaro, Pesaro, PU
  - UOC Chirurgia Generale - Ospedale "Regina Apostolorum" Albano Laziale (RM), Albano Laziale, RM
  - U.O. di Chirurgia Generale e d'Urgenza - Policlinico Casilino - Roma, Roma, RM
  - UOC Chirurgia Generale e Oncologica - Ospedale San Filippo Neri - ASL Roma1, Roma, RM
  - UOS Chirurgia Geriatrica - Policlinico Campus BioMedico - Roma, Roma, RM
  - UOC Chirurgia Generale, Laparoscopica, Toracica -Ospedale "Ceccarini" di Riccione - Area Vasta Romagna, Riccione, RN
  - UOC Chirurgia Generale 1 - Ospedale S. Chiara - APSS Trento, Trento, TN
  - UOC Chirurgia Generale - Ospedale "E. Agnelli" di Pinerolo (TO) - ASL TO3, Pinerolo, TO
  - UOC Chirurgia Generale - Ospedale Sacro Cuore Don Calabria Negrar Verona, Negrar, VR
  - UOC Chirurgia Generale Oncologica - Azienda Ospedaliera Belcolle - Viterbo, Viterbo, VT
  - SOC Chirurgia Colorettale - Istituto Nazionale dei Tumori - IRCCS Fondazione "G.Pascale" - Napoli, Napoli

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slieker JC, Komen N, Mannaerts GH, Karsten TM, Willemsen P, Murawska M, Jeekel J, Lange JF. Long-term and perioperative corticosteroids in anastomotic leakage: a prospective study of 259 left-sided colorectal anastomoses. Arch Surg. 2012 May;147(5):447-52. doi: 10.1001/archsurg.2011.1690. PMID 22249852
- [Background] Kingham TP, Pachter HL. Colonic anastomotic leak: risk factors, diagnosis, and treatment. J Am Coll Surg. 2009 Feb;208(2):269-78. doi: 10.1016/j.jamcollsurg.2008.10.015. Epub 2008 Dec 4. No abstract available. PMID 19228539
- [Background] Hyman N, Manchester TL, Osler T, Burns B, Cataldo PA. Anastomotic leaks after intestinal anastomosis: it's later than you think. Ann Surg. 2007 Feb;245(2):254-8. doi: 10.1097/01.sla.0000225083.27182.85. PMID 17245179
- [Background] Park JS, Choi GS, Kim SH, Kim HR, Kim NK, Lee KY, Kang SB, Kim JY, Lee KY, Kim BC, Bae BN, Son GM, Lee SI, Kang H. Multicenter analysis of risk factors for anastomotic leakage after laparoscopic rectal cancer excision: the Korean laparoscopic colorectal surgery study group. Ann Surg. 2013 Apr;257(4):665-71. doi: 10.1097/SLA.0b013e31827b8ed9. PMID 23333881
- [Background] Bruce J, Krukowski ZH, Al-Khairy G, Russell EM, Park KG. Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Br J Surg. 2001 Sep;88(9):1157-68. doi: 10.1046/j.0007-1323.2001.01829.x. PMID 11531861
- [Background] Lipska MA, Bissett IP, Parry BR, Merrie AE. Anastomotic leakage after lower gastrointestinal anastomosis: men are at a higher risk. ANZ J Surg. 2006 Jul;76(7):579-85. doi: 10.1111/j.1445-2197.2006.03780.x. PMID 16813622
- [Background] Platell C, Barwood N, Dorfmann G, Makin G. The incidence of anastomotic leaks in patients undergoing colorectal surgery. Colorectal Dis. 2007 Jan;9(1):71-9. doi: 10.1111/j.1463-1318.2006.01002.x. PMID 17181849
- [Background] Giaccaglia V, Salvi PF, Cunsolo GV, Sparagna A, Antonelli MS, Nigri G, Balducci G, Ziparo V. Procalcitonin, as an early biomarker of colorectal anastomotic leak, facilitates enhanced recovery after surgery. J Crit Care. 2014 Aug;29(4):528-32. doi: 10.1016/j.jcrc.2014.03.036. Epub 2014 Apr 5. PMID 24798346
- [Background] Ortega-Deballon P, Radais F, Facy O, d'Athis P, Masson D, Charles PE, Cheynel N, Favre JP, Rat P. C-reactive protein is an early predictor of septic complications after elective colorectal surgery. World J Surg. 2010 Apr;34(4):808-14. doi: 10.1007/s00268-009-0367-x. PMID 20049435
- [Background] Oberhofer D, Juras J, Pavicic AM, Rancic Zuric I, Rumenjak V. Comparison of C-reactive protein and procalcitonin as predictors of postoperative infectious complications after elective colorectal surgery. Croat Med J. 2012 Dec;53(6):612-9. doi: 10.3325/cmj.2012.53.612. PMID 23275327
- [Background] den Dulk M, Noter SL, Hendriks ER, Brouwers MA, van der Vlies CH, Oostenbroek RJ, Menon AG, Steup WH, van de Velde CJ. Improved diagnosis and treatment of anastomotic leakage after colorectal surgery. Eur J Surg Oncol. 2009 Apr;35(4):420-6. doi: 10.1016/j.ejso.2008.04.009. Epub 2008 Jun 27. PMID 18585889
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Skipper A, Ferguson M, Thompson K, Castellanos VH, Porcari J. Nutrition screening tools: an analysis of the evidence. JPEN J Parenter Enteral Nutr. 2012 May;36(3):292-8. doi: 10.1177/0148607111414023. Epub 2011 Nov 1. PMID 22045723
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Derived] Italian ColoRectal Anastomotic Leakage (iCral) study group; Borghi F, Migliore M, Cianflocca D, Ruffo G, Patriti A, Delrio P, Scatizzi M, Mancini S, Garulli G, Lucchi A, Carrara A, Pirozzi F, Scabini S, Liverani A, Baiocchi G, Campagnacci R, Muratore A, Longo G, Caricato M, Macarone Palmieri R, Vettoretto N, Ciano P, Benedetti M, Bertocchi E, Ceccaroni M, Pace U, Pandolfini L, Sagnotta A, Pirrera B, Alagna V, Martorelli G, Tirone G, Motter M, Sciuto A, Martino A, Scarinci A, Molfino S, Maurizi A, Marsanic P, Tomassini F, Santoni S, Capolupo GT, Amodio P, Arici E, Cicconi S, Marziali I, Guercioni G, Catarci M. Management and 1-year outcomes of anastomotic leakage after elective colorectal surgery. Int J Colorectal Dis. 2021 May;36(5):929-939. doi: 10.1007/s00384-020-03777-7. Epub 2020 Oct 29. PMID 33118101
- [Derived] Italian ColoRectal Anastomotic Leakage (iCral) study group. Risk factors for adverse events after elective colorectal surgery: beware of blood transfusions. Updates Surg. 2020 Sep;72(3):811-819. doi: 10.1007/s13304-020-00753-2. Epub 2020 May 12. PMID 32399595
- [Derived] Italian ColoRectal Anastomotic Leakage (iCral) Study Group. Anastomotic leakage after elective colorectal surgery: a prospective multicentre observational study on use of the Dutch leakage score, serum procalcitonin and serum C-reactive protein for diagnosis. BJS Open. 2020 Jun;4(3):499-507. doi: 10.1002/bjs5.50269. Epub 2020 Mar 5. PMID 32134216
- [Derived] Benedetti M, Ciano P, Pergolini I, Ciotti S, Guercioni G, Ruffo G, Borghi F, Patriti A, Del Rio P, Scatizzi M, Mancini S, Garulli G, Carrara A, Pirozzi F, Scabini S, Liverani A, Baiocchi G, Campagnacci R, Muratore A, Longo G, Caricato M, Macarone Palmieri R, Vettoretto N, Ceccaroni M, Guadagni S, Bertocchi E, Cianflocca D, Lambertini M, Pace U, Baraghini M, Pandolfini L, Angeloni R, Lucchi A, Martorelli G, Tirone G, Motter M, Sciuto A, Martino A, Luzzi AP, Di Cesare T, Molfino S, Maurizi A, Marsanic P, Tomassini F, Santoni S, Capolupo GT, Amodio P, Arici E, Clementi M, Ruggeri B, Catarci M. Early diagnosis of anastomotic leakage after colorectal surgery by the Dutch leakage score, serum procalcitonin and serum C-reactive protein: study protocol of a prospective multicentre observational study by the Italian ColoRectal Anastomotic Leakage (iC. G Chir. 2019 Jan-Feb;40(1):20-25. PMID 30771794
- [Derived] Italian ColoRectal Anastomotic Leakage (iCral) study group. Colorectal surgery in Italy: a snapshot from the iCral study group. Updates Surg. 2019 Jun;71(2):339-347. doi: 10.1007/s13304-018-00612-1. Epub 2019 Feb 11. PMID 30747374

DOCUMENTS (1):
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03560180/Prot_000.pdf